CLINICAL TRIAL: NCT01871025
Title: Early Incentive and Mobilization During COPD Exacerbation
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Diego Agustín Rodríguez, MD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/4025
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Hospitals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital and home exercise training (Experimental): Usual care plus hospital exercise training (aerobic and strength) followed by exercise training at home until 30 days to discharge.
  Interventions: Other: Hospital and home exercise training
- Usual care (Other): Usual care in COPD
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Hospital and home exercise training — Hospital exercise training (aerobic and strength) followed by exercise training
  Arms: Hospital and home exercise training
Other: Usual care — Usual care includes respiratory physiotherapy techniques during hospitalization and adequate physical activity recommendations, but not exercise training
  Other Names: Usual recommendations
  Arms: Usual care

SUMMARY:
To study the effects of early exercise training in hospitalized patients for Chronic Obstructive Pulmonary Disease exacerbation (COPD). Interventions are randomized. In one group, early exercise training (aerobic and strength) during hospitalization for COPD exacerbation followed by exercise training at home until 30 days to discharge and in the other the intervention is usual care. In both groups, usual respiratory physiotherapy techniques during hospitalization and adequate physical activity recommendations have been included. The main variable is the increase in moderate or vigorous daily physical activities at 30 days after discharge.

DETAILED DESCRIPTION:
Prospective randomized study in hospitalized patients for Chronic Obstructive Pulmonary Disease exacerbation (COPD). In one group, early exercise training (aerobic and strength) during hospitalization for COPD exacerbation followed by exercise training at home until 30 days to discharge and in the other the intervention is usual care. In both group, usual respiratory physiotherapy techniques during hospitalization and adequate physical activity recommendations have been included. The main variable is the increase in moderate or vigorous daily physical activities at 30 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients for COPD exacerbation

Exclusion Criteria:

* Hospitalization within the previous 14 days,
* current participation in rehabilitation program,
* locomotor or neurological condition or disability limiting the ability to perform exercise,
* lung transplantation or lung volume reduction surgery foreseen within 1 month after discharge.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Daily physical activity | 1 month
  Increase 10% moderate and/or vigorous daily physical activities after discharge

SECONDARY OUTCOMES:
Tolerance to exercise | 1 month
  Six minutes walk test
COPD Assessment Test (CAT) | 1 month
  Quality of life
Physical activity | 1 month
  International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Rodriguez, MD, Principal Investigator — Parc de Salut Mar
Locations (2):
- Spain (2):
  - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital Clinic i Provincial, Barcelona